CLINICAL TRIAL: NCT05206838
Title: Achilles Tendon Homograft for the Treatment of Gluteus Medius Insufficiency After Hip Replacement
Brief Title: Achilles Tendon for the Treatment of Gluteus Medius Insufficiency
Acronym: HLS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Göteborg University (Other); Vastra Gotaland Region (Other Government); The Swedish Society of Medicine (Other)
Responsible Party: Principal Investigator, Georgios Tsikandylakis, MD PhD, Senior consultant in orthopaedic surgery, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 276262
Record Dates: First submitted 2021-12-28; First posted 2022-01-25 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Arthroplasty Complications; Muscle Weakness; Muscle Atrophy; Muscle Tear
Keywords: Gluteus medius; Limp; Abductor; Trendelenburg
MeSH Terms: conditions — Muscle Weakness; Muscular Atrophy; Intermittent Claudication

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with the option of crossover in the control group after a certain period of time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Surgical reconstruction (Experimental): 22 patients undergo surgical reconstruction of gluteus medius with allograft consisting of Achilles tendon with calcaneus block. The calcaneus block is fixed into the greater trochanter and the Achilles tendon i passed through the gluteus medius muscle, tensioned and sutured into the muscle. Postoperatively, partial weight bearing for 2 months followed by physiotherapy for 10 months.
  Interventions: Procedure: Surgical reconstruction of gluteus medius with Achilles tendon allograft
- Physiotherapy (No Intervention): 22 patients receive non-operative treatment for their limp with physiotherapy alone during a 12-month period.

INTERVENTIONS:
Procedure: Surgical reconstruction of gluteus medius with Achilles tendon allograft — Achilles tendon allograft i fixed between the gluteus medius muscle and the greater trochanter
  Other Names: Homologous Achilles tendon transplant; Gastrocnemius tendon allograft
  Arms: Surgical reconstruction

SUMMARY:
Residual limping after total hip arthroplasty is a serious complication that lacks effective treatment. The purpose of this study is to evaluate a surgical treatment for residual limping and compare its results with non-surgical treatment. Our hypothesis is that surgical treatment followed by physiotherapy increases hip function and reduces limping compared with non-surgical treatment with physiotherapy alone.

DETAILED DESCRIPTION:
Residual limping due to gluteus medius insufficiency after total hip arthroplasty is a serious complication that lacks effective treatment. The purpose of this study is to evaluate surgical reconstruction of gluteus medius using Achilles tendon allograft and compare its results and adverse events with non-surgical treatment. Our hypothesis is that surgical reconstruction followed by physiotherapy increases hip function and reduces limping compared with non-surgical treatment with physiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Persisting limping with positive Trendelenburg's sign for at least 12 months after total hip arthroplasty
* Rupture/avulsion of the gluteus medius tendon verified with ultrasound or MRI
* Leg length discrepancy of less than 1 cm
* Femoral offset discrepancy of less than 25%

Exclusion Criteria:

* Neuromuscular disorders

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Oxford Hip Score (OHS) | 12 months
  Patient-reported hip function measured in a scale 0-48

SECONDARY OUTCOMES:
Trendelenburg's sign | 12 months
  Presence or abscence of Trendelenburg's sign as binary outcome (yes/no)
Hip abduction torque | 12 months
  Abduction torque in the frontal plane measured in Nm/Kg with gait analysis
University of California Level of Activity (UCLA) | 12 months
  Patient-reported activity level measured with in a rank scale 0-10
Euroqol 5 dimension 5 level index (EQ5D-5L) | 12 months
  Patient-reported health-related quality of life measured with swedish version of the euroqol 5 dimension 5 level index in a scale 0-1
Euroqol visual analog scale (EQVAS) | 12 months
  Patient-reported health-related quality of life measured with the euroqol visual analog scale 0-100
Adverse events | 12 months
  All complications resulting in contact with health care provider within one year.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Tsikandylakis, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whiteside LA, Roy ME. Incidence and treatment of abductor deficiency during total hip arthroplasty using the posterior approach: repair with direct suture technique and gluteus maximus flap transfer. Bone Joint J. 2019 Jun;101-B(6_Supple_B):116-122. doi: 10.1302/0301-620X.101B6.BJJ-2018-1511.R1. PMID 31146555
- [Background] Ewen AM, Stewart S, St Clair Gibson A, Kashyap SN, Caplan N. Post-operative gait analysis in total hip replacement patients-a review of current literature and meta-analysis. Gait Posture. 2012 May;36(1):1-6. doi: 10.1016/j.gaitpost.2011.12.024. Epub 2012 Mar 10. PMID 22410129
- [Background] Whiteside LA. Surgical technique: Transfer of the anterior portion of the gluteus maximus muscle for abductor deficiency of the hip. Clin Orthop Relat Res. 2012 Feb;470(2):503-10. doi: 10.1007/s11999-011-1975-y. PMID 21796476
- [Background] Fehm MN, Huddleston JI, Burke DW, Geller JA, Malchau H. Repair of a deficient abductor mechanism with Achilles tendon allograft after total hip replacement. J Bone Joint Surg Am. 2010 Oct 6;92(13):2305-11. doi: 10.2106/JBJS.I.01011. PMID 20926725
- [Background] Beard DJ, Harris K, Dawson J, Doll H, Murray DW, Carr AJ, Price AJ. Meaningful changes for the Oxford hip and knee scores after joint replacement surgery. J Clin Epidemiol. 2015 Jan;68(1):73-9. doi: 10.1016/j.jclinepi.2014.08.009. Epub 2014 Oct 31. PMID 25441700